CLINICAL TRIAL: NCT01892904
Title: A Multi-center, Randomized, Open-label, Active-controlled, Parallel-group Comparative Study to Assess Efficacy and Safety of a Flexible Extended Regimen of BAY 86-5300 (0.02 mg Ethinylestradiol [β-CDC] and 3 mg Drospirenone) Compared to the 28-day (24 + 4-day) Regimen of BAY 86-5300 in the Treatment of Dysmenorrhea for 24 Weeks
Brief Title: Comparative Study of BAY86-5300 With a Flexible Extended Regimen for Dysmenorrhea
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16114
Record Dates: First submitted 2013-07-02; First posted 2013-07-08 (Estimated); Last update posted 2015-09-09 (Estimated); Status verified 2015-09

CONDITIONS: Dysmenorrhea
Keywords: YAZ; Flexible regimen; Drospirenone; Ethinylestradiol Betadex; Dysmenorrhea; Japanese patients
MeSH Terms: conditions — Dysmenorrhea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- EE20/DRSP(BAY86-5300)-flexibel extended regimen (Experimental): One tablet [0.02 mg of ethinylestradiol (β-CDC) and 3 mg of drospirenone] / day with flexible extended regimen (24-day to 120-day active tablet intake followed by 4-day tablet free interval)
  Interventions: Drug: EE20/DRSP(BAY86-5300)
- EE20/DRSP(BAY86-5300)-28 days cyclic regimen (Active Comparator): One tablet [0.02 mg of ethinylestradiol (β-CDC) and 3 mg of drospirenone] / day with 28-day cyclic regimen (24-day active tablet intake followed by 4-day placebo tablet intake)
  Interventions: Drug: EE20/DRSP(BAY86-5300)

INTERVENTIONS:
Drug: EE20/DRSP(BAY86-5300) — One tablet [0.02 mg of ethinylestradiol (β-CDC) and 3 mg of drospirenone] / day

SUMMARY:
The is a multi-center, randomized, open-label, active-controlled, parallel-group comparative study (24-week treatment period).

The objective of this study is to prove the superiority of BAY 86-5300 with flexible extended regimen for treatment of dysmenorrhea to BAY 86-5300 with 28-day cyclic regimen in terms of primary efficacy variable, number of days with dysmenorrheic pain over 140 days of evaluation period.

In addition, the long-term safety of the flexible extended regimen of BAY86-5300 in patients treated for one year will be investigated.

ELIGIBILITY:
Inclusion Criteria: - Dysmenorrhea patients with a total dysmenorrhea score (sum of the two sub-scores: severity of dysmenorrhea and use of analgesics) of at least 3 points in each of the last two menstruations before randomization (baseline observation phase)

* Patients with dysmenorrheic pain during the 2 baseline cycles before randomization. Dysmenorrheic pain means any spasmodic pelvic pain or lower abdominal pain with possible radiation towards back or thighs recorded in the Patient Diary in correspondence with a withdrawal and/or menstrual bleeding episode. Pain could start up to 2 days before the onset of the bleeding episode the bleeding and terminates on the last day of bleeding of before
* Patients having the regular cyclic menstrual period (25 to 38 days) in the latest two menses before randomization (baseline observation phase)
* Willingness to use a barrier method (i.e., non-hormonal method) for contraception during the study. Acceptable methods of contraception include (i) condoms (male or female) with or without a spermicidal agent; (ii) diaphragm or cervical cap with spermicide; (iii) intra-uterine device.

Exclusion Criteria: - Patients who have organic diseases of which surgical treatment is prioritized by the investigator

* Patients aged 40 years or older with ovarian chocolate cysts being more than 10 cm in size of the longest diameters
* Patients with ovarian chocolate cysts having solid part in the cyst
* Patients for whom YAZ Combination Tablet is contraindicated (according to Japanese Labeling)

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Actual)
Dates: Start 2013-07; Primary Completion 2015-01 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Number of days with dysmenorrheic pain over 140 days of evaluation period | Evaluation period which starts on 25th day after start of treatment and lasts for 140 days
  Number of days with dysmenorrheic pain is determined based on daily record of Patient Diary.

SECONDARY OUTCOMES:
Change in Dysmenorrhea score from baseline to period of withdrawal bleeding | Baseline period (8 weeks before start of treatment) and evaluation period which starts on 25th day after start of treatment and lasts for 140 days
  Dysmenorrhea score is a sum of the two sub-scores, severity of dysmenorrhea and use of analgesics, recorded by the participant at every visit
Change of severity of pain Description | Baseline period (8 weeks before start of treatment) and evaluation period which starts on 25th day after start of treatment and lasts for 140 days
  The severity of pain is measured by the Visual Analogue Scale (VAS), recorded by the participant at any visit.
Number of days with at least moderate dysmenorrheic pain over 140 days of evaluation period | Evaluation period which starts on 25th day after start of treatment and lasts for 140 days
  Number of days with at least moderate dysmenorrheic pain is determined based on daily record of Patient Diary.
Number of days with rescue medicine used for relief of dysmenorrhea or pelvic pain over 140 days of evaluation period | Evaluation period which starts on 25th day after start of treatment and lasts for 140 days
  Number of days with rescue medicine is determined based on daily record of Patient Diary.
Number of days with interference of dysmenorrheic pain with daily activity over 140 days of evaluation period | Evaluation period which starts on 25th day after start of treatment and lasts for 140 days
  Number of days with interference of dysmenorrheic pain with daily activity is determined based on daily record of Patient Diary
Endometrial thickness | 24 weeks after taking the initial study medication
  Endometrial thickness is the thickest value (mm) of endometrium determined by transvaginal ultrasonography.
Number of days with bleeding and spotting over treatment phase | Up to 24 weeks
  Number of days with spotting/bleeding is determined based on daily record of Patient Diary.

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (7):
- Japan (7):
  - Matsudo, Chiba
  - Osaka, Osaka
  - Hachiōji, Tokyo
  - Minato, Tokyo
  - Setagaya-ku, Tokyo
  - Suginami-ku, Tokyo
  - Toshima-ku, Tokyo

REFERENCES:
- [Derived] Momoeda M, Akiyama S, Yamamoto S, Kondo M, Fukai T. Burden of Menstrual Pain Measured by Heatmap Visualization of Daily Patient-Reported Data in Japanese Patients Treated with Ethinylestradiol/Drospirenone: A Randomized Controlled Study. Int J Womens Health. 2020 Mar 10;12:175-185. doi: 10.2147/IJWH.S242864. eCollection 2020. PMID 32210639